CLINICAL TRIAL: NCT01239862
Title: Phase-1 Study of Autologous Bone Marrow Cells Intrabronchial Instillation for Patients Silicosis
Brief Title: Safety of Stem Cells Intrabronchial Instillation for Silicosis
Acronym: SilicStemCell
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); Ministry of Health, Brazil (Other Government); National Research Council, Brazil (Other)
Responsible Party: Principal Investigator, Marcelo Marcos Morales, MD, PhD, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONEP5772008
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic and Accelerated Silicosis
Keywords: pulmonary, silicosis, chronic and accelerated silicosis, autologous transplantation; bone marrow cells, stem cells, cell therapy
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Silicosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous cell transplantation (Experimental): We conducted a prospective, non-randomized, single-center longitudinal study in five patients. Inclusion criteria were age 18-50 years, chronic and accelerated silicosis, forced expiratory volume in 1s <60% and >40%, forced vital capacity ≥60% and arterial oxygen saturation >90%. BMDMCs were administered through bronchoscopy (2×107 cells) into both lungs. Physical examination, laboratory evaluations, quality of life questionnaires, thoracic computed tomography scans, lung function tests, and perfusion scintigraphy were performed before the beginning of treatment and up to 360 days after BMDMC (Bone Marrow Derived Mononuclear Cells) therapy. Additionally, whole-body and planar scans were evaluated 2 and 24 h after instillation.
  Interventions: Other: Autologous cell transplantation

INTERVENTIONS:
Other: Autologous cell transplantation — Intrabronchial Instillation Of Bone Marrow Derived Mononuclear Cells

SUMMARY:
The aim of this study was to analyze the safety, pulmonary function, and quality of life data of patients with silicosis treated with intrabronchial instillation of bone marrow derived mononuclear cells (BMDMC, 2x107) through bronchoscopy.

DETAILED DESCRIPTION:
This study will perfume the safety (Phase I) study of 10 patients with silicosis treated with intrabronchial instillation of autologous bone marrow derived mononuclear cells (BMDMC, 2x107) through bronchoscopy. The inclusion criteria is: age between 18-50, chronic and accelerated silicosis, characterized with a fibrotic increase in the last two years, FEV1 <60% and > 40%, FVC > 60% and SaO2 >90%, while the exclusion criteria were: smoking, active tuberculosis or other infections, cancer, auto-immune disorders, hematological, hepatic or cardiac diseases, and pregnancy. All patients will be subjected to clinical examination, answered questionnaires of quality of life (SGRQ and SF36) and dyspnea score (Borg), performed high resolution CT of thorax, pulmonary function tests with DLCO and 6-minute walk test and lung perfusion scintigraphy before and 7, 30, 60, 180 and 360 days after treatment.

For each patient, 2×107 cells will be labeled with 99mTc. Briefly, 500 μl of sterile SnCl2 solution is added to the cells and the mixture is incubated at room temperature for 10 min. Forty-five mCi of 99mTc is then added and incubation continued for another 10 min. After centrifugation (500×g for 5 min), the supernatant is removed and the cells are washed in saline solution. The pellet was also resuspended in saline solution. Viability of the labeled cells was assessed by the trypan blue exclusion test, and was estimated to be greater than 93% in all cases. Labeling efficiency (%) was calculated by the activity in the pellet divided by the sum of the radioactivity in the pellet plus supernatant and was estimated to be greater than 90% in all cases. Whole body and planar scans will be performed 2 and 24h after instillation. Perfusion scintigraphy will be performed before and 30, 60, 120 and 180 days after BMDMC therapy. For regional analysis the right and left lungs will be divided into three zones: base, midzone, and apex.

ELIGIBILITY:
Inclusion Criteria:age between 18-50, chronic and accelerated silicosis, characterized with a fibrotic increase in the last two years, FEV1 <60% and > 40%, FVC > 60% and SaO2 >90%

Exclusion Criteria: smoking, active tuberculosis or other infections, cancer, auto-immune disorders, hematological, hepatic or cardiac diseases, and pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Absence of lung deficits during the procedure and/or in the 4 months follow-up | 4 months

SECONDARY OUTCOMES:
Improvement of pulmonary deficits | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Clementino Fraga Filho - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Morales MM, Souza SA, Loivos LP, Lima MA, Szklo A, Vairo L, Brunswick TH, Gutfilen B, Lopes-Pacheco M, Araujo AJ, Cardoso AP, Goldenberg RC, Rocco PR, Fonseca LM, Lapa e Silva JR. Pilot safety study of intrabronchial instillation of bone marrow-derived mononuclear cells in patients with silicosis. BMC Pulm Med. 2015 Jun 11;15:66. doi: 10.1186/s12890-015-0061-8. PMID 26059242